CLINICAL TRIAL: NCT01571167
Title: A Human Laboratory Assessment of the Safety and Potential Efficacy of Varenicline in Methamphetamine-Dependent Volunteers Receiving Methamphetamine
Brief Title: Varenicline as a Treatment for Methamphetamine Dependence
Acronym: Varenicline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard De La Garza, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: H-26875; DPMC (Other: NIDA); 1R01DA027134-01 (NIH)
Record Dates: First submitted 2012-02-20; First posted 2012-04-05 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Methamphetamine Dependence; Methamphetamine Abuse; Substance Abuse
Keywords: Methamphetamine; Chantix; Varenicline
MeSH Terms: conditions — Substance-Related Disorders | interventions — Sugars; Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Varenicline 2 mg (Active Comparator)
  Interventions: Drug: Varenicline
- Varenicline 1 mg (Active Comparator)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Placebo — Participants will receive varenicline or matched placebo from day 1 through day 7, then the same subjects will return within 2-4 weeks and assigned to each of the two remaining study medication conditions, and undergo the identical procedures (3-phase study).
  Other Names: Sugar pill
  Arms: Placebo
Drug: Varenicline — For varenicline 1 mg, dosing will begin at 0.5 mg once daily (with 0 mg placebo to maintain blind of bid dosing) for days 1-3, will be increased to 0.5 mg twice daily for the days 4-6, and then reduced to 0.5 mg once daily on day 7. No medication is given on Day 8.
  Other Names: Chantix
  Arms: Varenicline 1 mg
Drug: Varenicline — For varenicline 2 mg, dosing will begin at 0.5 mg once daily for days 1-3 (with 0 mg placebo to maintain blind of bid dosing), will be increased to 0.5 mg twice daily for day 4, and increased to 1 mg twice daily on days 5-6, and then reduced to 1 mg once daily on day 7. No medication is given on Day 8.
  Other Names: Chantix
  Arms: Varenicline 2 mg

SUMMARY:
The primary purpose of the study is to determine the effects of treatment with varenicline (1 and 2 mg daily), compared to treatment with placebo, on methamphetamine-induced craving and subjective effects in methamphetamine-dependent human volunteers.

DETAILED DESCRIPTION:
This study is part of an effort to develop treatments for methamphetamine abuse. Varenicline is a drug that changes levels of certain brain chemicals that may also be useful in helping people to stop using methamphetamine. Our goal is to determine the safety and effects of varenicline (1 and 2 mg, daily, vs. a placebo) when it is used before experimental administration of methamphetamine, on a number of physical and psychological measures; specifically blood pressure, heart rate, and how you feel after taking methamphetamine. The secondary purpose is to determine the effects of treatment with varenicline (1 and 2 mg daily), compared to treatment with placebo, on the reinforcing effects of methamphetamine by measuring methamphetamine self-administration in methamphetamine-dependent human volunteers.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in the study, participants must:

1. Be English-speaking volunteers who are not seeking treatment at the time of the study
2. Be between 18-55 years of age
3. Meet DSM-IV TR criteria for MA dependence
4. Must be cigarette smokers, defined as smoking 10 or more cigarettes per day by self-report
5. Have a self-reported history of using MA by the smoked or IV route and provide at least one MA-positive urine prior to admission
6. Have vital signs as follows: resting pulse between 50 and 90 bpm, blood pressures between 105-150 mm Hg systolic and 45-90 mm Hg diastolic; this criterion must be met within 2 days of admission
7. Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal
8. Have a baseline EKG that demonstrates normal sinus rhythm, normal conduction (including QTc), and no clinically significant arrhythmias
9. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician or nurse practitioner and the principal investigator.

Exclusion Criteria:

Subjects will be excluded if they:

1. Have any previous medically adverse reaction to METH, including loss of consciousness, chest pain, or epileptic seizure
2. Have neurological or psychiatric disorders, as assessed by MINI, such as: episode of major depression within the past 2 years; lifetime history of schizophrenia, other psychotic illness, or bipolar illness; current organic brain disease or dementia assessed by clinical interview; history of or any current psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; history of suicide attempts within the past three months and/or current suicidal ideation/plan; history of psychosis occurring in the absence of current METH use
3. Meet DSM-IV criteria for abuse/dependence on alcohol or other drugs, except nicotine or marijuana
4. Have used methamphetamine only by the intravenous route
5. Have evidence of clinically significant heart disease or hypertension, as determined by physician
6. Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
7. Have HIV and currently symptomatic, have a diagnosis of AIDS, or currently taking antiretroviral medication
8. Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, and throughout the study
9. Have any history of asthma, chronic coughing and wheezing, or other chronic respiratory illnesses
10. Currently use alpha or beta agonists, theophylline, or other sympathomimetics
11. Have made a suicide attempt in the past year
12. Have any other illness, condition, or use of medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of study.

Criteria for Discontinuation Following Initiation:

1. Positive urine drug screen or breath test indicating illicit use of cocaine, MA, alcohol, opiates, or other abused drugs not delivered as part of this protocol
2. Inability to comply with study procedures
3. Meet discontinuation criteria due to exaggerated response to MA, described below
4. Nausea severe enough to require treatment.

Rationale for Subject Selection Criteria:

Participants are required to have used MA by the smoked or IV route to avoid exposing participants to routes of administration that produce more intensive interoceptive effects. The age criteria were selected primarily to avoid enrolling participants with undiagnosed cardiovascular disease. Participants with active HIV disease are excluded to avoid potential exacerbation of their underlying disease; participants with asymptomatic HIV are included because this group is at high risk for MA dependence. Participants with asthma (or who take asthma medications) are excluded due to potential adverse interactions between beta agonist medications and MA.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The effects of varenicline and methamphetamine on safety and cardiovascular measures | On study day 6 and 7
  The safety of MA administration during treatment will be assessed by reporting of adverse events (AEs), and using ECG recording, and heart rate and blood pressure measurements. Digital 12-lead ECG will also be recorded prior to randomization. Blood pressure and heart rate will be measured from 15 min prior to MA or placebo dosing until 2 h after dosing. In addition, heart rate and blood pressure will be assessed throughout the inpatient portion of the protocol.

SECONDARY OUTCOMES:
The effects of varenicline and methamphetamine on subjective effects | On study day 6 and 7
  Efficacy will be assessed by measuring effects of treatment on subjective effects produced by administration of MA. Patients will complete visual analog scale (VAS) ratings at T= 5, 15, 30, 60, 120, 240 and 360 min post dosing. Other diagnostic measures and assessment instruments will be used to further characterize the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Richard De La Garza, II, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kalechstein AD, Mahoney JJ 3rd, Verrico CD, De La Garza R 2nd. Short-term, low-dose varenicline administration enhances information processing speed in methamphetamine-dependent users. Neuropharmacology. 2014 Oct;85:493-8. doi: 10.1016/j.neuropharm.2014.05.045. Epub 2014 Jun 12. PMID 24930359
- [Derived] Verrico CD, Mahoney JJ 3rd, Thompson-Lake DG, Bennett RS, Newton TF, De La Garza R 2nd. Safety and efficacy of varenicline to reduce positive subjective effects produced by methamphetamine in methamphetamine-dependent volunteers. Int J Neuropsychopharmacol. 2014 Feb;17(2):223-33. doi: 10.1017/S146114571300134X. PMID 24393456